CLINICAL TRIAL: NCT03645473
Title: Evaluation of Device Settings for Airway Clearance Using The Monarch Airway Clearance System
Acronym: HFCWO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CR-RR-2018-002
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Monarch device settings assessment group (Experimental): Patients with cystic fibrosis who have experience with the Monarch Airway Clearance System will be enrolled in the study.
  The duration of subject participation is approximately 4 - 6 hours during 1 study visit. Each subject will receive therapy with The Monarch® System at multiple frequency and intensity combinations as defined in the Study procedures.
  Interventions: Device: Monarch Airway Clearance System

INTERVENTIONS:
Device: Monarch Airway Clearance System — HFCWO Airway Clearance Device

SUMMARY:
The study will be an open label laboratory study with all subjects receiving HFCWO with The Monarch® System

Objective:

Assess device settings and to identify frequency/pressure (intensity) combinations that produce high airflow and oscillating volume

Methodology:

Subjects will receive HFCWO using The Monarch® System at multiple frequency / intensity combinations on a single visit day. Frequency / intensity combinations will be evaluated to determine which settings produce highest airflow and highest oscillating volume.

DETAILED DESCRIPTION:
The study will be an open-label, laboratory study. All enrolled subjects will receive HFCWO therapy with the Monarch® system. The study will be conducted at one (1) site in the US.

The study will evaluate oscillating airflow and oscillating volume induced during therapy with the Monarch® system. Subjects will also rate the comfort of the therapy. Patients with cystic fibrosis (CF) who meet all of the inclusion criteria and none of the exclusion criteria will be enrolled in the study.

Therapy with the Monarch® system will be delivered using multiple frequency/intensity combination settings. The order of settings will be randomized for each study subject. During therapy oscillating flow and volume measurements will be obtained for each frequency/intensity combination. Following each frequency/intensity combination, subjects will respond to a subjective assessment of the comfort of the therapy by rating the comfort on a visual analogue scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF (by sweat test and/or genetics
* Age > 15 years
* Require regular home airway clearance therapy
* Current user of The Monarch® System with a minimum of 4 weeks experience with the device
* Signed informed consent. If patient is a minor, parents/guardians must give written informed consent and patient must give written assent
* Patient must be on a stable regimen of CF medication

Exclusion Criteria:

* History of pneumothorax within the past 6 months prior to study visit
* History of hemoptysis requiring embolization within the past 12 months prior to study visit or hemoptysis of > 100 ml within a 24-hour period within the past 30 days
* History of lobectomy
* Recent chest surgery or chest trauma
* Inability to perform The Monarch® System therapy as directed
* Pregnant or lactating female
* Have a pacemaker or implantable cardioverter defibrillator (ICD)
* Requirement for oral or IV antibiotics that are not part of the subject's usual course of treatment within the past 14 days prior to screening

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-01-24 (Estimated); Primary Completion 2019-03-12 (Estimated); Study Completion 2019-04-12 (Estimated)

PRIMARY OUTCOMES:
Peak oscillating expiratory airflow measurements | 4-6 hours
  Subjects will be treated with the Monarch® system using multiple frequency/intensity combination settings. After adjusting the therapy to the desired setting, subjects will be instructed breath through the mouthpiece for the flow measurement system, to breathe normally and continue relaxed breathing. Oscillating flow and volume measurement will be captured by the system over a period of 30 to 60 seconds of relaxed breathing.
  Data from the measurement of oscillating flow for each frequency/intensity combination setting will be processed following the completion of the testing

SECONDARY OUTCOMES:
Oscillating volume | 4-6 hours
  Oscillating volume measurement will be conducted concurrently with the measurement of flow. Subjects will be treated with the Monarch® system using multiple frequency/intensity combination settings as described above.
  Data from the measurement of oscillating volume for each frequency/intensity combination setting will be processed following the completion of the testing
Patient comfort/discomfort evaluated by 100 mm visual analogue scale (VAS) | 4-6 hours
  Following the completion of testing for each frequency/intensity combination setting, subjects will rate the level of comfort/discomfort of the setting on a VAS.
  A Visual Analogue Scale is a psychometric response scale which will be used as a measuring instrument for subjective comfort or discomfort. It is a measurement instrument that ranges across a continuum of values and used to measure the intensity or frequency of various symptoms.
  * The Visual Analogue Scale ranges from (0 to 100 mm).
  * Zero means very uncomfortable/intolerable and 100 means very comfortable.
  The subject will mark the line for each setting combination to indicate the level of comfort or discomfort.
  After the Study visit, the research staff will measure the mark on the line and document the value.